CLINICAL TRIAL: NCT05180604
Title: Improving Patients With Chronic Disease to Engage in the eHealth Care Environment: the Application and Evaluation of eHealth Literacy Concept
Brief Title: The Application and Evaluation of eHealth Literacy (eHL) Concept
Acronym: eHL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yu-Chi Chen, Associate professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MOST-107-2314-B-010-014-MY3
Record Dates: First submitted 2021-11-15; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Kidney Diseases; Cardiovascular Diseases
Keywords: Chronic disease; eHealth literacy; patient engagement; experience learning theory; Self-management; empowerment; eHealth care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Cardiovascular Diseases; Chronic Disease; Patient Participation; Empowerment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experience learning programs of eHealth care (Experimental): Patients in the experimental group received 6 sections of activities.
  Interventions: Behavioral: experience learning programs of eHealth care
- Usual care (No Intervention): Patients in control group received usual care

INTERVENTIONS:
Behavioral: experience learning programs of eHealth care — The experience learning programs of eHealth care was included six sections of activities. Six activities were conducted based on eHealth literacy framework and experience learning theory to improve patients' abilities to engage in eHealth care service. The outcome indicators were eHealth literacy, patient health engagement, the acceptance of eHealth care, eHealth usage status, and their learning experience
  Arms: experience learning programs of eHealth care

SUMMARY:
This study aims to explore the effectiveness of experience learning program of eHealth care to improve the chronic patients' eHL in engaging with the eHealth care system on the indicators on eHealth literacy, patient health engagement, e-Health usage status among Chronic disease patients included type 2 diabetes patients, Chronic kidney disease, and Cardiovascular Diseases.

DETAILED DESCRIPTION:
Chronic diseases are irreversible that incurs considerable medical and economic costs. Even if the government and medical health care system make an effort to improve care and recommend e-health care, the incidence and prevalence rates of chronic diseases have not decreased but increased, and participants have even become the main cause of kidney disease. Technology and daily life has become more inseparable, which also led to the change of the traditional face to face health care model. The chronic disease care is gradually transitioning into the smart eHealth care era, patients are in need of learning how to face innovative ways of using care and resources. eHealth literacy (eHL)is the essential element that determines if patient can adapt to the rapidly changing health care system.

Due to the disciplinary integration of medical and technology, eHealth care provides continuous care for patients. But, it is still necessary to return to patient-centered care thinking and improving patients' knowledge and ability to use eHealth care technology. This can be applied to disease care, and implemented for daily self-health management. Therefore, this study explores the effects of intervention and the learning process and experience of patients through an experience learning program of eHealth care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as a type 2 diabetes patients, Chronic kidney disease, and Cardiovascular Diseases more than three months.
* At least 20 years old, with clear consciousness and able to communicate in Mandarin or Taiwanese.
* Possess a mobile phone or tablet with internet capabilities.
* Consent to participate in this research and be willing to sign a consent form.

Exclusion Criteria:

* Suffering from serious diseases, such as: general paralysis, mental disorders, cognitive function abnormalities, etc.
* Those who cannot communicate in Mandarin or Taiwanese.
* Those who refuse to participate in this research.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Baseline of eHealth Literacy Questionnaire scores | The pretest is completed when the patients agrees to join the intervention.
  Evaluate the patient's eHL level, including 7 dimensions (1) Using technology to process health information, (2) Understanding of health concepts and languages, (3)Ability to actively engage with digital service, (4)Feel safe and in control, (5) Motivated to engage with digital service, (6) Access to digital services that work (7)Digital services that suit individual. The higher the score, the better the eHL.
The eHealth Literacy Questionnaire scores at the end of intervention | The post-test 1 is completed at the end of the 6 weeks intervention
  Evaluate the patient's eHL level, including 7 dimensions (1) Using technology to process health information, (2) Understanding of health concepts and languages, (3)Ability to actively engage with digital service, (4)Feel safe and in control, (5) Motivated to engage with digital service, (6) Access to digital services that work (7)Digital services that suit individual. The higher the score, the better the eHL.
The eHealth Literacy Questionnaire scores after intervention at 3 months | The post-test 2 is completed after intervention at 3 months
  Evaluate the patient's eHL level, including 7 dimensions (1) Using technology to process health information, (2) Understanding of health concepts and languages, (3)Ability to actively engage with digital service, (4)Feel safe and in control, (5) Motivated to engage with digital service, (6) Access to digital services that work (7)Digital services that suit individual. The higher the score, the better the eHL.
The eHealth Literacy Questionnaire scores after intervention at 6 months | The post-test 3 is completed after intervention at 6 months
  Evaluate the patient's eHL level, including 7 dimensions (1) Using technology to process health information, (2) Understanding of health concepts and languages, (3)Ability to actively engage with digital service, (4)Feel safe and in control, (5) Motivated to engage with digital service, (6) Access to digital services that work (7)Digital services that suit individual. The higher the score, the better the eHL.
Baseline of The acceptance of eHealth care scores | The pretest is completed when the patients agrees to join the intervention.
  The scale was developed base on Technology Acceptance Model to assess patients' behaviors intention of using the eHealth device
The acceptance of eHealth care scores at the end of intervention | The post-test 1 is completed at the end of the 6 weeks intervention
  The scale was developed base on Technology Acceptance Model to assess patients' behaviors intention of using the eHealth device
The acceptance of eHealth care scores after intervention at 3 months | The post-test 2 is completed after intervention at 3 months
  The scale was developed base on Technology Acceptance Model to assess patients' behaviors intention of using the eHealth device
The acceptance of eHealth care scores after intervention at 6 months | The post-test 3 is completed after intervention at 6 months
  The scale was developed base on Technology Acceptance Model to assess patients' behaviors intention of using the eHealth device
Baseline of Health Technology Usage Sore | The pretest is completed when the patients agrees to join the intervention.
  Use self-developed structured questionnaires to investigate the types of health technology use and monitoring items. Use types include computer or network systems, mobile apps, health monitoring systems or wearable devices (such as pedometers, smart bracelets, heart rate monitors, blood pressure monitors, Blood glucose meter, blood pressure meter, blood glucose meter or weight scale, etc.) or other, monitoring items include blood pressure, blood sugar, weight, diet, sleep, heart rate, steps or other health data. The higher the number, the more items are monitored, the total score The higher the level, the better the use of health technology.
The Health Technology Usage Sore at the end of intervention | The post-test 1 is completed at the end of the 6 weeks intervention
  Use self-developed structured questionnaires to investigate the types of health technology use and monitoring items. Use types include computer or network systems, mobile apps, health monitoring systems or wearable devices (such as pedometers, smart bracelets, heart rate monitors, blood pressure monitors, Blood glucose meter, blood pressure meter, blood glucose meter or weight scale, etc.) or other, monitoring items include blood pressure, blood sugar, weight, diet, sleep, heart rate, steps or other health data. The higher the number, the more items are monitored, the total score The higher the level, the better the use of health technology.
The Health Technology Usage Sore after intervention at 3 months | The post-test 2 is completed after intervention at 3 months
  Use self-developed structured questionnaires to investigate the types of health technology use and monitoring items. Use types include computer or network systems, mobile apps, health monitoring systems or wearable devices (such as pedometers, smart bracelets, heart rate monitors, blood pressure monitors, Blood glucose meter, blood pressure meter, blood glucose meter or weight scale, etc.) or other, monitoring items include blood pressure, blood sugar, weight, diet, sleep, heart rate, steps or other health data. The higher the number, the more items are monitored, the total score The higher the level, the better the use of health technology.
The Health Technology Usage Sore after intervention at 6 months | The post-test 3 is completed after intervention at 6 months
  Use self-developed structured questionnaires to investigate the types of health technology use and monitoring items. Use types include computer or network systems, mobile apps, health monitoring systems or wearable devices (such as pedometers, smart bracelets, heart rate monitors, blood pressure monitors, Blood glucose meter, blood pressure meter, blood glucose meter or weight scale, etc.) or other, monitoring items include blood pressure, blood sugar, weight, diet, sleep, heart rate, steps or other health data. The higher the number, the more items are monitored, the total score The higher the level, the better the use of health technology.
Baseline of Patient Health Engagement score | The pretest is completed when the patients agrees to join the intervention.
  The scale is thought of as a self-administering tool by the patient in order to diagnose his/ her This scale has a total of 5 questions. The higher the number, the higher the patient engagement it is.
The Patient Health Engagement score at the end of the intervention | The post-test 1 is completed at the end of the 6 weeks intervention
  The scale is thought of as a self-administering tool by the patient in order to diagnose his/ her This scale has a total of 5 questions. The higher the number, the higher the patient engagement it is.
The Patient Health Engagement score after intervention at 3 months | The post-test 2 is completed after intervention at 3 months
  The scale is thought of as a self-administering tool by the patient in order to diagnose his/ her This scale has a total of 5 questions. The higher the number, the higher the patient engagement it is.
The Patient Health Engagement score after intervention at 6 months | The post-test 3 is completed after intervention at 6 months
  The scale is thought of as a self-administering tool by the patient in order to diagnose his/ her This scale has a total of 5 questions. The higher the number, the higher the patient engagement it is.

SECONDARY OUTCOMES:
The change in renal function level at the end of the intervention | To collect two-time point data by chart review. Those were before the intervention and the end of the the 6 weeks intervention
  The health outcome indicator of management of renal disease by using the estimated Glomerular filtration rate(eGRF) .
The change Trajectory of renal function level from baseline to after intervention at 6 months and 1 year | To collect three-time point data by chart review. Those were before the intervention, the end of the 6 weeks intervention, and after intervention at six months and 1 year
  The health outcome indicator of management of renal disease by using the estimated Glomerular filtration rate(eGRF) .
The change in HbA1C level at the end of the intervention | To collect two-time point data by chart review. Those were before the intervention and the end of the the 6 weeks intervention
  The health outcome indicator of management of diabetes
The change Trajectory of HbA1C level from baseline to after the intervention at 3, 6, and 12 months | To collect four-time point data by chart review. Those were before the intervention, the end of the 6 weeks intervention, after the intervention at three months, after the intervention at six months, and after the intervention at twelve months
  The health outcome indicator of management of diabetes
The change in Triglycerides level at the end of the intervention | To collect two-time point data by chart review. Those were before the intervention and the end of the six weeks intervention
  The health outcome indicator of management of lipid
The change Trajectory of Triglycerides level from baseline to after the intervention at 3 , 6 and 12 months | To collect four-time point data by chart review. Those were before the intervention, the end of the 6 weeks intervention, after the intervention at three months, after the intervention at six months, and after the intervention at twelve months.
  The health outcome indicator of management of lipid
The change in Cholesterol level at the end of the intervention | To collect two-time point data by chart review. Those were before the intervention and the end of the 6 weeks intervention
  The health outcome indicator of management of lipid
The change Trajectory of Cholesterol level from baseline to after the intervention at 3, 6 and 12 months | To collect two-time point data by chart review. Those were before the intervention, the end of the 6 weeks intervention, after the intervention at three months, after the intervention at six months, and after the intervention at twelve months.
  The health outcome indicator of management of lipid

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chi Chen, Ph.D., Study Chair — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kayser L, Karnoe A, Furstrand D, Batterham R, Christensen KB, Elsworth G, Osborne RH. A Multidimensional Tool Based on the eHealth Literacy Framework: Development and Initial Validity Testing of the eHealth Literacy Questionnaire (eHLQ). J Med Internet Res. 2018 Feb 12;20(2):e36. doi: 10.2196/jmir.8371. PMID 29434011
- [Result] Graffigna G, Barello S, Bonanomi A, Lozza E. Measuring patient engagement: development and psychometric properties of the Patient Health Engagement (PHE) Scale. Front Psychol. 2015 Mar 27;6:274. doi: 10.3389/fpsyg.2015.00274. eCollection 2015. PMID 25870566
- [Result] Kayser L, Kushniruk A, Osborne RH, Norgaard O, Turner P. Enhancing the Effectiveness of Consumer-Focused Health Information Technology Systems Through eHealth Literacy: A Framework for Understanding Users' Needs. JMIR Hum Factors. 2015 May 20;2(1):e9. doi: 10.2196/humanfactors.3696. PMID 27025228
- [Result] Richtering SS, Morris R, Soh SE, Barker A, Bampi F, Neubeck L, Coorey G, Mulley J, Chalmers J, Usherwood T, Peiris D, Chow CK, Redfern J. Examination of an eHealth literacy scale and a health literacy scale in a population with moderate to high cardiovascular risk: Rasch analyses. PLoS One. 2017 Apr 27;12(4):e0175372. doi: 10.1371/journal.pone.0175372. eCollection 2017. PMID 28448497
- [Result] Schillinger D. The Intersections Between Social Determinants of Health, Health Literacy, and Health Disparities. Stud Health Technol Inform. 2020 Jun 25;269:22-41. doi: 10.3233/SHTI200020. PMID 32593981
- [Result] Alpay L, van der Boog P, Dumaij A. An empowerment-based approach to developing innovative e-health tools for self-management. Health Informatics J. 2011 Dec;17(4):247-55. doi: 10.1177/1460458211420089. PMID 22193825
- [Result] Knight E, Stuckey MI, Petrella RJ. Health promotion through primary care: enhancing self-management with activity prescription and mHealth. Phys Sportsmed. 2014 Sep;42(3):90-9. doi: 10.3810/psm.2014.09.2080. PMID 25295771
- [Result] Kreps GL, Neuhauser L. New directions in eHealth communication: opportunities and challenges. Patient Educ Couns. 2010 Mar;78(3):329-36. doi: 10.1016/j.pec.2010.01.013. Epub 2010 Mar 3. PMID 20202779
- [Derived] Cheng YS, Lin CP, Chen LA, Hwang WR, Lin YC, Chen YC. Short-Term Effects of an eHealth Care Experiential Learning Program Among Patients With Type 2 Diabetes: Randomized Controlled Trial. J Med Internet Res. 2024 Aug 16;26:e53509. doi: 10.2196/53509. PMID 39150761
- See also: A Multidimensional Tool Based on the eHealth Literacy Framework: Development and Initial Validity Testing of the eHealth Literacy Questionnaire (eHLQ) — https://doi.org/10.2196/jmir.8371
- See also: Measuring patient engagement: development and psychometric properties of the Patient Health Engagement (PHE) Scale. — https://doi.org/10.3389/fpsyg.2015.00274